CLINICAL TRIAL: NCT07362121
Title: Assessment of the Verus Frame as a Support for the Leg in Orthopaedic Surgery (Intramedullary Nailing) of Tibial Fracture in Adults. A Prospective, Single-arm, Interventional Post-market Clinical Investigation With AO Foundation Approved Acceptance Criteria and a Retrospective Registry Control Group.
Brief Title: Assessment of the Verus Frame in Tibial Intramedullary Nailing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hemitec Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VERUS-001_PMCFSP
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verus_patients (Experimental): Verus is intended to be used as a support of leg during orthopaedic surgery. The post-operative alignment and rotation will be determined by x-ray and computed tomography scan.
  Interventions: Device: Verus frame to stabilize tibia

INTERVENTIONS:
Device: Verus frame to stabilize tibia — Verus is used during tibial intramedullary nailing surgery.

SUMMARY:
This prospective, single-arm Post-Market Clinical Follow-Up (PMCF) study, utilizing a registry-based control group, will assess the Verus frame's effectiveness in achieving precise tibial rotation and alignment during intramedullary nailing procedure, as well as safety of the device. The results will be compared to AO-approved criteria to ensure comprehensive evaluation of its new benefits, regulatory compliance, and continued clinical use. Tibial intramedullary nailing is the gold standard for tibial fracture fixation, where accurate alignment and rotation are crucial for optimal recovery and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Tibial fracture to be operated by suprapatellar intramedullary nailing technique
* 18-80 years old
* Signed informed consent

Exclusion Criteria:

* Situations where intramedullary fixation is otherwise contraindicated, e.g., active or potential infection, osteoporosis or where a patient's cooperation cannot be guaranteed.
* Pregnancy, breastfeeding
* Open fractures with severe soft tissue damage
* Polytrauma
* Previous tibia fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Post-operative X-ray measurement of alignment | Within two days after operation
  Varus/valgus alignment measurement and anterior/posterior angulation measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland